CLINICAL TRIAL: NCT06397560
Title: PrOton Pulsed reduCed dOse Rate Radiotherapy for Recurrent CNS maligNancies (POPCORN) Trial
Brief Title: PrOton Pulsed reduCed dOse Rate Radiotherapy for Recurrent CNS maligNancies Trial
Acronym: POPCORN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Ion Beam Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KOT-001
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-03

CONDITIONS: Glioma; Glioma, Malignant; Recurrent Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRDR Radiotherapy (Experimental)
  Interventions: Radiation: PRDR

INTERVENTIONS:
Radiation: PRDR — Proton pulsed reduced dose rate (PRDR) technique, to a dose of 54 Gy in 30 fractions (treatments) with proton radiotherapy. Treatments will occur once per day on consecutive weekdays.

SUMMARY:
The purpose of this research study is to see if a specific type of radiation therapy, called "proton pulsed reduced dose rate" or "PRDR radiotherapy" has any benefits at dose levels and number of fractions thought to be acceptable in earlier research studies. The researchers want to find out what effects (good and bad) PRDR has on people with cancer in the brain called a "recurrent high-grade glioma" meaning that it grows fast, can spread quickly, and it has come back or gotten worse after being treated previously.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status ≥ 50
* Histologically-confirmed or radiographic evidence of recurrent / progressive glioma
* Prior treatment with radiotherapy to a minimum dose of 45 Gy
* At least 6 months or greater between completion of prior radiotherapy and enrollment in this study. If prospective participants have not passed an interval of at least 6 months, they may still be eligible if they meet one or more of the following criteria:

  1. New areas of tumor outside the original radiotherapy fields as determined by the investigator.
  2. Histologic confirmation of tumor through biopsy or resection AND an interval of at least 90 days between completion of radiotherapy and enrollment.
  3. Nuclear medicine imaging, magnetic resonance (MR) spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than radiation necrosis obtained within 28 days of enrollment AND an interval of at least 90 days between completion of radiotherapy and enrollment.
* Must have recovered from grade 3+ toxicities of prior therapy and there must be a minimum time of 28 days prior to enrollment from the administration of any investigational agent or prior cytotoxic therapy
* Must not be pregnant (positive pregnancy test) or breastfeeding. Must agree to use of highly effective contraception during radiotherapy treatment and for an additional 6 months. Should a participant become pregnant or suspect that they are pregnant while participating in this study, they should notify the treating physician immediately.

Highly effective and acceptable forms of contraception are:

* Male condom plus spermicide
* Cap plus spermicide
* Diaphragm plus spermicide
* Copper T
* Progesterone T
* Levonorgestrel-releasing intrauterine system (e.g., Mirena®)
* Implants
* Hormone shot or injection
* Combined pill
* Mini-pill
* Patch

Individuals who meet any of the following criteria will not need contraception:

* Individuals assigned male at birth
* Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments
* Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the postmenopausal range for individuals under 50
* Radiation-induced oophorectomy with last menses > 1 year ago
* Chemotherapy-induced menopause with >1 year interval since last menses
* Surgical sterilization (bilateral oophorectomy or hysterectomy)

Exclusion Criteria:

* Two or more courses of prior radiotherapy
* Inability to undergo an MRI with contrast
* Leptomeningeal evidence of recurrent disease
* Multi-focal disease
* Any other condition that may put a participant at higher risk, at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 3 months
  PFS is defined as the duration of time from treatment start to first progressive disease (PD), date of death, or last follow-up date on which the patient was reported alive after proton PRDR reirradiation. Response to treatment will be assessed using Response Assessment in Neuro-Oncology (RANO).

SECONDARY OUTCOMES:
Treatment-related adverse events (AEs) assessed by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) | 2 years
  The total number of AEs considered possibly, probably, or definitely related to proton PRDR as per the CTCAE v5.0.
Overall survival (OS) | 2 years
  OS is defined as the duration of time from treatment start to date of death, or last follow-up date on which the patient was reported alive after proton PRDR reirradiation.
Grade 3 central nervous system (CNS) toxicities assessed by CTCAE v5.0 | 2 years
  The number of CNS AEs considered possibly, probably, or definitely related to proton PRDR as per CTCAE v5.0
Assessment of symptoms using the MD Anderson Symptom Inventory for Brain Tumors (MDASI-BT) | 1 year
  Symptoms will be assessed using the MDASI-BT, which is a 28-item questionnaire that asks about cancer symptoms and how the symptoms interfere with daily life. Each item is scored on a 0-10 scale (0 = best, 10 = worst), with a total score of 0-280, with a higher score indicating worse symptoms.
Quality of life (QOL) assessed by the EuroQOL 5-dimension, 5-level (EQ-5D-5L) | 1 year
  QOL will be assessed using the EQ-5D-5L questionnaire. There are five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. There also is a visual analog scale asking about overall health that ranges from 0-100. Higher scores indicate better health and QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Press, M.D., Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (2):
- United States (2):
  - Lynn Cancer Institute at Baptist Health, Inc., Boca Raton, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adkison JB, Tome W, Seo S, Richards GM, Robins HI, Rassmussen K, Welsh JS, Mahler PA, Howard SP. Reirradiation of large-volume recurrent glioma with pulsed reduced-dose-rate radiotherapy. Int J Radiat Oncol Biol Phys. 2011 Mar 1;79(3):835-41. doi: 10.1016/j.ijrobp.2009.11.058. Epub 2010 May 14. PMID 20472350
- [Background] Bovi JA, Prah MA, Retzlaff AA, Schmainda KM, Connelly JM, Rand SD, Marszalkowski CS, Mueller WM, Siker ML, Schultz CJ. Pulsed Reduced Dose Rate Radiotherapy in Conjunction With Bevacizumab or Bevacizumab Alone in Recurrent High-grade Glioma: Survival Outcomes. Int J Radiat Oncol Biol Phys. 2020 Nov 15;108(4):979-986. doi: 10.1016/j.ijrobp.2020.06.020. Epub 2020 Jun 27. PMID 32599030
- [Background] Dilworth JT, Krueger SA, Dabjan M, Grills IS, Torma J, Wilson GD, Marples B. Pulsed low-dose irradiation of orthotopic glioblastoma multiforme (GBM) in a pre-clinical model: effects on vascularization and tumor control. Radiother Oncol. 2013 Jul;108(1):149-54. doi: 10.1016/j.radonc.2013.05.022. Epub 2013 Jun 19. PMID 23791366
- [Background] Kotecha R, Odia Y, Khosla AA, Ahluwalia MS. Key Clinical Principles in the Management of Glioblastoma. JCO Oncol Pract. 2023 Apr;19(4):180-189. doi: 10.1200/OP.22.00476. Epub 2023 Jan 13. PMID 36638331
- [Background] Kutuk T, Tolakanahalli R, McAllister NC, Hall MD, Tom MC, Rubens M, Appel H, Gutierrez AN, Odia Y, Mohler A, Ahluwalia MS, Mehta MP, Kotecha R. Pulsed-Reduced Dose Rate (PRDR) Radiotherapy for Recurrent Primary Central Nervous System Malignancies: Dosimetric and Clinical Results. Cancers (Basel). 2022 Jun 15;14(12):2946. doi: 10.3390/cancers14122946. PMID 35740612
- [Background] Saeed AM, Khairnar R, Sharma AM, Larson GL, Tsai HK, Wang CJ, Halasz LM, Chinnaiyan P, Vargas CE, Mishra MV. Clinical Outcomes in Patients with Recurrent Glioblastoma Treated with Proton Beam Therapy Reirradiation: Analysis of the Multi-Institutional Proton Collaborative Group Registry. Adv Radiat Oncol. 2020 Apr 22;5(5):978-983. doi: 10.1016/j.adro.2020.03.022. eCollection 2020 Sep-Oct. PMID 33083661
- See also: Baptist Health Cancer Care — https://baptisthealth.net/services/cancer-care